CLINICAL TRIAL: NCT04082611
Title: The PREVENTION Trial: Precision Recommendations for Environmental Variables, Exercise, Nutrition and Training Interventions to Optimize Neurocognition
Brief Title: The PREVENTION Trial: Precision Recommendations to Optimize Neurocognition
Acronym: PREVENTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint John's Cancer Institute (Other)
Collaborators: Institute for Systems Biology (Other); St. Joseph's Healthcare Foundation (Other)
Responsible Party: Principal Investigator, David Merrill, Associate Professor, Department of Translational Neurosciences & Neurotherapeutics; Director, Pacific Brain Health Center, Saint John's Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20190583
Record Dates: First submitted 2019-07-24; First posted 2019-09-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Alzheimer Disease; Mild Cognitive Impairment; Precision Medicine; Health Coaching; Multi-Modal Intervention; Personal, Dense, Dynamic Data (PD3) Clouds; Cognitive decline
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be assigned with a participant identification number (ID), so that data will not be identified by any names or personally identifiable information. This ID will be used throughout this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Data-driven clinical recommendations (CR) (Active Comparator): Data-driven clinical recommendations (CR)
  Interventions: Behavioral: Data-Driven Clinical Recommendations
- Group 2 - Data-driven coached multi-modal intervention (MMIC) (Experimental): Data-driven coached multi-modal intervention (MMIC)
  Interventions: Behavioral: Coached Data-Driven Clinical Recommendations

INTERVENTIONS:
Behavioral: Data-Driven Clinical Recommendations — Data-driven clinical recommendations. Participants will receive routine care with data-driven, personalized, multi-modal clinical recommendations by a study physician based on study assessments and clinical lab values and be monitored and re-assessed for a period of 12 months.
  Arms: Group 1 - Data-driven clinical recommendations (CR)
Behavioral: Coached Data-Driven Clinical Recommendations — Data-driven multi-modal lifestyle intervention with coaching. Participants will receive coached routine care with data-driven, personalized, multimodal recommendations. MMIC participants will receive an intensive multi-modal intervention with health coaching, support and resources to carry out these recommendations. This additional intervention services include: 13 personal, data-driven brain health coaching sessions (with an RDN), 7 personal dietary counseling sessions (with an RDN), 33 group-based cognitive and physical exercise classes (CogFit) with a certified personal trainer and a computer-based neurocognitive program at home and be monitored and re-assessed for a period of 12 months.
  Arms: Group 2 - Data-driven coached multi-modal intervention (MMIC)

SUMMARY:
The PREVENTION Trial is a 12-month, two-arm randomized clinical trial (RCT) in adults 50-80 years old experiencing cognitive decline. Our study clinicians will refer patients for enrollment based on three categories: 1) a diagnosis of mild AD according to criteria established by the National Institute of Neurological and Communicative Disorders and Stroke (AD and Related Disorders Association [NINCDS-ADRDA]), 2) those with mild cognitive impairment will be diagnosed according to the Petersen method, and 3) subjective memory impairment as assessed by neuropsychological assessments and self-report. Enrollment will require evidence of AD pathophysiological processes (as defined by a positive amyloid positron emission tomography (PET) scan).

The first objective is to evaluate the efficacy of a coached, data-driven, multi-modal lifestyle intervention to treat cognitive decline. Subjects will be randomized into one of two groups: Group 1 (Active Control) or Group 2 (Intervention). Group 1 (Data-driven clinical recommendations (CR)) will serve as the active control group and will receive data-driven clinical recommendations by a study physician based on study assessments and clinical lab values. Group 2 (Data-driven multi-modal intervention with coaching (MMIC)) will receive the same clinical recommendations and also an intensive multi-modal intervention with health coaching, support and resources to carry out these recommendations. This includes health coaching sessions (with an RDN), dietary counseling sessions (with an RDN), and group cognitive and physical exercise classes (CogFit) with a certified personal trainer and a computer-based neurocognitive program at home. Both groups will be measured for treatment related changes in cognitive and functional abilities, quality of life, biological, and biochemical measures.

The second objective is to analyze longitudinal multi-omic data, including metabolomics, proteomics, genetics, microbiome, behavior and cognition into personalized, dense, dynamic data (i.e. PD3) from individuals with cognitive decline and underlying Alzheimer's neuropathology. The goal analysis is to identify models of causation that can further advance knowledge and research in neurodegenerative disorders and healthy living.

DETAILED DESCRIPTION:
Subject identification and recruitment - All participants will be recruited from the Pacific Brain Health Center in Santa Monica, which is a high-volume memory-care and dementia outpatient clinic within a large physician medical group affiliated with Providence Saint John's Health Center. 60 participants will be randomized into the RCT, with 30 in each treatment arm.

Procedures for Obtaining Informed Consent - All participants will receive the Experimental Research Subject's Bill of Rights prior to signing the informed consent form (ICF), authorization of use and disclosure of protected health information (PHI), and authorization of medical record release for the subject's treating physician, will be obtained from each participants prior to enrolling in the study. A copy of all signed ICF's will be given to the participants, and the investigator will retain the original.

A Functional Assessment Staging Test (FAST) will be done before participants are consented to determine whether they or a legally appointed representative (LAR) can consent to participate in the study. In this study, participants with FAST stages 2-4 will be recruited (see Inclusion Criteria).

Considerations for consenting: FAST Stages 2-3 Participants - FAST stages 2-3 participants are usually capable of making medical and legal decisions, and will be consented directly, unless there is a caregiver, legally appointed representative, or other reason to think that an informed consent cannot be given by the participants without approval by a reliable informant acting on their behalf.

Considerations for consenting: FAST Stage 4 (mild dementia) Participants - FAST stage 4 participants will be consented by having them give oral or written assent, indicating their preference with regard to study participation. In addition, the caregiver or legally appointed representative of a demented participants will be consented to assure full understanding of study procedures and willingness on behalf of the participants to participate in the study.

The consenting approach for patients with cognitive impairment has been evaluated by the Department of Psychiatry and Behavioral Sciences at Johns Hopkins, and found to adequately ensure informed consent. They concluded that ADRD participants should not be excluded from study participation if they cannot directly consent themselves, so long as their caregivers can consent, and the participants can assent, either verbally or in writing, their preference to participate in the study.

The caregiver or legally appointed representative will be required to accompany participants to participate in the required procedures. A copy of the appropriate document (e.g., the power of attorney for healthcare) will be obtained and filed with the original ICF.

ELIGIBILITY:
Inclusion Criteria

* Subjects must be age 50 to 80 at time of informed consent.
* Subjects of any gender, race or ethnicity are eligible to enroll in the study.
* Subjects must have a FAST stage of 2-4.
* Subjects with FAST Stage 4 must have a caregiver or legally appointed representative willing to accompany participants to the required procedures.
* As part of the study screening procedure, subjects must be willing to undergo an amyloid PET scan or have previously undergone an amyloid PET scan and agree to make the results available. Subjects must be amyloid positive to be eligible to enroll in the study.
* Subjects must be proficient in spoken and written English for consenting as well as for study participation since the intervention in this study (e.g., coaching program) is currently only available in English.
* Subjects with medical conditions must be stable for these conditions. Stable control on medication is acceptable. Subjects should not have started any new medications for chronic conditions within the last three months.
* A neurological and physical evaluation will be conducted prior to enrollment of the study by a qualified medical doctor and confirmed through medical records that they do not possess any abnormal physical or neurological sign, and/ whether they are considered to be clinically significant. Also an MMSE >19 will be confirmed by a medical doctor prior to study enrollment.
* Subjects, with or without assistance, must be able to use a computer and web interface. If assistance is needed, it must be readily available to them.
* Subjects must be able to converse with a coach telephonically. Video-based telephone coaching is part of data-driven health coaching.
* Subjects must have regular access to a computer and the Internet along with dedicated email address since certain aspects of the program (e.g. cognitive training) are delivered electronically.
* Subject must have normal visual acuity (or corrected to normal) and normal color vision as indicated by self-report.
* Subject must have adequate hearing acuity as indicated by self-report.
* Subject must have adequate motor capacity to use a mobile phone/iPad/computer as indicated by self-report and confirmed by staff before they are enrolled into a treatment arm.
* Subject must be cleared by a physician to participate in a moderately intensive exercise program.

Exclusion Criteria

* Subjects with an existing diagnosis of a non-AD neurodegenerative disorder (e.g., Lewy Body Dementia, Frontal-Temporal Dementia).
* Subjects with a diagnosis of cerebrovascular disease as the primary cause of cognitive impairment.
* A previously reported AD high-risk mutation (e.g., in the Presenilin Protein (PSEN) or Amyloid Precursor Protein (APP) genes) in the participant or immediate family (children, siblings, or parents). Such patients may accumulate amyloid faster than in late onset AD, and therefore may show less pronounced benefit from intervention.
* Mini Mental State Exam (MMSE) below 20.
* Clinical Dementia Rating (CDR) global score of 2 or above.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
NIH ToolBox Cognition Function Battery - Cognitive Function Composite Score | 1 year
  To test the hypothesis that high contact coaching is better than no coaching for people in the early stages and at risk for cognitive decline. We plan to test that after one year of coached data-driven personalized interventions, participants in the coaching (CDDCR) (Group 2) will have less cognitive decline than the non-coaching (DDCR) arm (Group 1) as measured by the NIH ToolBox Cognition Function Battery (NIHTB-CB).
  The Cognitive Function Composite Score will be our primary outcome measure for cognitive function. The NIHTB-CB contains seven computer-based instruments assessing five cognitive sub-domains: Language, Executive Function, Episodic Memory, Processing Speed, and Working Memory. The Composite Score is calculated using all seven subsets of the NIHTB-CB. Participants will be assessed at baseline and one year.
RAVLT (Rey's Auditory Verbal Learning Test) score | 1 year
  To test the hypothesis that high contact coaching is better than no coaching for people in the early stages and at risk for cognitive decline. We plan to test that after one year of coached data-driven personalized interventions, participants in the coaching (CDDCR) (Group 2) will have less cognitive decline than the non-coaching (DDCR) arm (Group 1) as measured by the he Rey Auditory Verbal Learning Test (RAVLT). The RAVLT is a test derived for assessing verbal learning and memory. The RAVLT will be used to evaluate the changes in memory function of participants in the two different arms. Participants will be assessed at baseline and one year. Changes in RAVLT learn and recall scores will be used to assess changes in cognitive function.
Hippocampal Volume | 1 year
  To test the hypothesis that high contact coaching is better than no coaching for people in the early stages and at risk for cognitive decline. We plan to test that after one year of coached data-driven personalized interventions, participants in the coaching (CDDCR) (Group 2) will have less hippocampal volume decline than the non-coaching (DDCR) arm (Group 1) as measured by the structural magnetic resonance imaging (MRI). Participants will be assessed at baseline and one year.

SECONDARY OUTCOMES:
Blood Urine Nitrogen | 1 year
  To test the hypothesis that high contact coaching is better than no coaching for people in the early stages and at risk for cognitive decline. We plan to test that after one year of coached data-driven personalized interventions, participants in the coaching (CDDCR) (Group 2) will have lower blood urea levels (BUN) than the non-coaching (DDCR) arm (Group 1) as measured by the plasma BUN. Participants will be assessed at baseline and one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific Brain Health Center, Santa Monica, California, United States

REFERENCES:
- [Background] Barnes DE, Yaffe K. The projected effect of risk factor reduction on Alzheimer's disease prevalence. Lancet Neurol. 2011 Sep;10(9):819-28. doi: 10.1016/S1474-4422(11)70072-2. Epub 2011 Jul 19. PMID 21775213
- [Background] Lidman D, Ek AC, Dahllof AG, Eldh J, Palmer B, Hultling C. [Bedsores--etiology, prevention and treatment]. Lakartidningen. 1989 Nov 8;86(45):3880-2. No abstract available. Swedish. PMID 2811536
- [Background] Friedenreich CM, Courneya KS, Bryant HE. The lifetime total physical activity questionnaire: development and reliability. Med Sci Sports Exerc. 1998 Feb;30(2):266-74. doi: 10.1097/00005768-199802000-00015. PMID 9502356
- [Background] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Background] Park YH, Moon SH, Ha JY, Lee MH. The long-term effects of the health coaching self-management program for nursing-home residents. Clin Interv Aging. 2017 Jul 11;12:1079-1088. doi: 10.2147/CIA.S137821. eCollection 2017. PMID 28744111
- [Background] Jack CR Jr, Bernstein MA, Fox NC, Thompson P, Alexander G, Harvey D, Borowski B, Britson PJ, L Whitwell J, Ward C, Dale AM, Felmlee JP, Gunter JL, Hill DL, Killiany R, Schuff N, Fox-Bosetti S, Lin C, Studholme C, DeCarli CS, Krueger G, Ward HA, Metzger GJ, Scott KT, Mallozzi R, Blezek D, Levy J, Debbins JP, Fleisher AS, Albert M, Green R, Bartzokis G, Glover G, Mugler J, Weiner MW. The Alzheimer's Disease Neuroimaging Initiative (ADNI): MRI methods. J Magn Reson Imaging. 2008 Apr;27(4):685-91. doi: 10.1002/jmri.21049. PMID 18302232
- [Background] Pfeffer RI, Kurosaki TT, Harrah CH Jr, Chance JM, Filos S. Measurement of functional activities in older adults in the community. J Gerontol. 1982 May;37(3):323-9. doi: 10.1093/geronj/37.3.323. PMID 7069156
- [Background] Price ND, Magis AT, Earls JC, Glusman G, Levy R, Lausted C, McDonald DT, Kusebauch U, Moss CL, Zhou Y, Qin S, Moritz RL, Brogaard K, Omenn GS, Lovejoy JC, Hood L. A wellness study of 108 individuals using personal, dense, dynamic data clouds. Nat Biotechnol. 2017 Aug;35(8):747-756. doi: 10.1038/nbt.3870. Epub 2017 Jul 17. PMID 28714965
- [Background] Thom DH, Hessler D, Willard-Grace R, DeVore D, Prado C, Bodenheimer T, Chen EH. Health coaching by medical assistants improves patients' chronic care experience. Am J Manag Care. 2015 Oct;21(10):685-91. PMID 26633093
- [Background] Willard-Grace R, Chen EH, Hessler D, DeVore D, Prado C, Bodenheimer T, Thom DH. Health coaching by medical assistants to improve control of diabetes, hypertension, and hyperlipidemia in low-income patients: a randomized controlled trial. Ann Fam Med. 2015 Mar;13(2):130-8. doi: 10.1370/afm.1768. PMID 25755034
- [Background] Norton S, Matthews FE, Barnes DE, Yaffe K, Brayne C. Potential for primary prevention of Alzheimer's disease: an analysis of population-based data. Lancet Neurol. 2014 Aug;13(8):788-94. doi: 10.1016/S1474-4422(14)70136-X. PMID 25030513
- [Background] Slavich GM, Shields GS. Assessing Lifetime Stress Exposure Using the Stress and Adversity Inventory for Adults (Adult STRAIN): An Overview and Initial Validation. Psychosom Med. 2018 Jan;80(1):17-27. doi: 10.1097/PSY.0000000000000534. PMID 29016550
- [Background] Washburn RA, McAuley E, Katula J, Mihalko SL, Boileau RA. The physical activity scale for the elderly (PASE): evidence for validity. J Clin Epidemiol. 1999 Jul;52(7):643-51. doi: 10.1016/s0895-4356(99)00049-9. PMID 10391658
- [Background] Hansmannel F, Sillaire A, Kamboh MI, Lendon C, Pasquier F, Hannequin D, Laumet G, Mounier A, Ayral AM, DeKosky ST, Hauw JJ, Berr C, Mann D, Amouyel P, Campion D, Lambert JC. Is the urea cycle involved in Alzheimer's disease? J Alzheimers Dis. 2010;21(3):1013-21. doi: 10.3233/JAD-2010-100630. PMID 20693631
- [Background] McKhann G, Drachman D, Folstein M, Katzman R, Price D, Stadlan EM. Clinical diagnosis of Alzheimer's disease: report of the NINCDS-ADRDA Work Group under the auspices of Department of Health and Human Services Task Force on Alzheimer's Disease. Neurology. 1984 Jul;34(7):939-44. doi: 10.1212/wnl.34.7.939. PMID 6610841
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol. 1999 Mar;56(3):303-8. doi: 10.1001/archneur.56.3.303. PMID 10190820
- See also: Jacobs, P. (Ed.). (2017). NSCA's Essentials of Training Special Populations. Human Kinetics. — https://books.google.com/books?id=8DAtDwAAQBAJ&pg=PA459&lpg=PA459&dq=Jacobs,+P.+(Ed.).+(2017).+NSCA%27s+Essentials+of+Training+Special+Populations.+Human+Kinetics.&source=bl&ots=xfOeLBhO-N&sig=ACfU3U3rj-6QOloF2EuMVf0X3Wm7QZp8Fw&hl=en&sa=X&ved=2ahUKEwiE_8r07bnjAhWD_J4KHTP7BR0Q6AEwBnoECAkQAQ#v=onepage&q=Jacobs%2C%20P.%20(Ed.).%20(2017).%20NSCA's%20Essentials%20of%20Training%20Special%20Populations.%20Human%20Kinetics.&f=false